CLINICAL TRIAL: NCT06468046
Title: Mama Empoderada: Adapting a Novel Mental Health Prevention Intervention for Migrant Mothers With Young Children in a Humanitarian Setting
Brief Title: Mama Empoderada: Adapting a Novel Mental Health Prevention Intervention for Migrant Mothers With Young Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: El Colegio de la Frontera Norte (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-2023-0135
Record Dates: First submitted 2024-06-10; First posted 2024-06-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Interventional
Keywords: parenting intervention; mental health; migrant mothers
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The pilot randomized controlled trial (RCT) of the adapted 'Mama Empoderada' intervention with Migrant Mothers will include N=100 [N(treatment)=50; N(control)=50] (Aims 2-3). The intervention group (IG) will participate in trauma- informed group and individual sessions addressing parenting, active linkage to resources, social support, and resilience. The control group will receive standard of care programming, including referrals to drop-in migrant and community-based supports, childcare, and referrals to reproductive, mental health, and other services. Control group participants will have the opportunity to participate in the full intervention following completion of the intervention and all questionnaires by the intervention group (post 6-month visit). Both groups will complete baseline, exit, and follow-up (2, 4, 6-months) surveys.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mama Empoderada (Mom Power) (Experimental): Behavioral: The intervention group will receive the Mama Empoderada intervention, which is a theory- based, trauma-informed, culturally tailored group intervention to promote mental health and positive parenting outcomes among trauma-exposed mothers with young children (0-5 years). Intervention participants will receive 10 group and 3 individual sessions addressing parenting, active linkage to resources (e.g., food, shelter, migration), social support, and resilience.
  Interventions: Behavioral: Mama Empoderada [Mom Power]
- Standard of care (No Intervention): The control group will receive standard of care programming available locally, including referrals to drop-in migrant and family supports, childcare, and referrals to reproductive, mental health, and other services. Control group participants will have the opportunity to participate in the full intervention following completion of the intervention and all questionnaires by the intervention group (post 6-month visit).

INTERVENTIONS:
Behavioral: Mama Empoderada [Mom Power] — 'Mamá Empoderada' [Mom Power] is a theory-based, trauma-informed group intervention to promote mental health and positive parenting among mothers with young children (0-5 years). It has been adapted for migrant mothers, and will conduct a pilot randomized controlled trial (RCT) of the intervention with migrant mothers with young children (MMC). The intervention group (IG) will receive 10 group and 3 individual sessions addressing attachment theory, hands-on parenting skills, linkage to resources (e.g., food, shelter), social support, and self-care and resilience.
  Arms: Mama Empoderada (Mom Power)

SUMMARY:
This pilot randomized controlled trial will test a theory-based, trauma-informed, and culturally-tailored intervention [Mama Empoderada' (Mom Power)] to promote mental health and positive parenting among migrant mothers with young children.

DETAILED DESCRIPTION:
The goal of this randomized controlled trial is to adapt and pilot-test a novel mental health prevention intervention for migrant mothers with young children in a humanitarian setting.

This pilot trial will adapt 'Mama Empoderada' [Mom Power] - a theory-based, trauma-informed, culturally-tailored group intervention to promote mental health and positive parenting among mothers with young children (0-5 years) for the first time. Aims are to:

1. Conduct a pilot study of the adapted intervention to determine acceptability and estimate effect sizes on symptoms of depression, anxiety, and parenting stress; and
2. Explore which theory-based mechanisms of action predict changes in symptoms of depression, anxiety, and parenting stress, and identify factors associated with differential intervention response.

The intervention group will receive trauma-informed group and individual sessions on parenting, linkage to resources (e.g., food, shelter), social support, and resilience. The control group will receive standard of care programming.

Both groups will complete baseline and exit surveys, as well as follow-up surveys at 2-, 4- and 6- months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a mother to at least one accompanying child <6 years of age
* At least 18 years old
* Migrated to Tijuana from a Latin American country other than Mexico, or born in Mexico and internally displaced
* Able to provide informed consent
* Screen below cut-offs for major depression and anxiety disorder
* Able to speak Spanish
* Available to participate in full duration of 'Mama Empoderada'

Exclusion Criteria

* Not a mother or only accompanied by older children (> age 6)
* Less than 18 years of age
* Migrated to Tijuana from region outside of Latin America or non-migrant
* Unable to provide informed consent
* Screen above cut-offs for major depression and anxiety disorders
* Unable to speak Spanish
* Unable to participate in full intervention (either control or intervention group).

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms (Patient Health Questionnaire [PHQ]-9) | Baseline, post-intervention (Approximately 6-weeks after baseline), and post-intervention follow-ups (2-months, 4-months, and 6-months post-intervention)
  Survey of Depression symptoms (PHQ-9), scores range from 1-27 with higher scores indicating more severe depression
Anxiety symptoms (General Anxiety Disorder [GAD]-7) | baseline, post-intervention (approximately 6-weeks after baseline), and post-intervention follow-up (2-months, 4-months, and 6-months post-intervention)
  Survey of Anxiety symptoms (GAD-7), scores range from 0-21, with higher scores indicating higher levels of anxiety.
Parental Stress Scale | baseline, post-intervention (approximately 6-weeks after baseline), and post-intervention follow-up (2-months, 4-months, and 6-months post-intervention)
  Survey of Parental Stress, Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.

CONTACTS AND LOCATIONS:
Overall Officials: Shira Goldenberg, PhD, Principal Investigator — San Diego State University
Locations (1):
- Al Otro Lado, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
NIMH requires data that involve human subjects to be shared using the NDA (see NOT-MH-23-100). Quantitative data from this pilot trial will be preserved to enable sharing via NDA data of sufficient quality to validate and replicate research findings described in the Aims as noted below.

REFERENCES:
- [Derived] Goldenberg SM, Ramage K, Martinez-Torteya C, Pitpitan E, Rosenblum K, Hernandez C, Alvarez M, Rangel G, Bojorquez-Chapela I. Mama Empoderada: study protocol for a pilot trial of a novel parenting and mental health prevention intervention for migrant mothers with young children at the Mexico-US border. BMJ Open. 2025 Jan 28;15(1):e094917. doi: 10.1136/bmjopen-2024-094917. PMID 39880445